CLINICAL TRIAL: NCT04886115
Title: Effects of Eccentric Pedaling at Different Rates on Neuromuscular Function
Acronym: Exo-Mode 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LAROCHE 2021
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Volunteers Who Can do Moderate Physical Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric pedalling group at 15 rpm (Experimental)
  Interventions: Other: Neuromuscular evaluation; Other: Assessment of aerobic capacity, muscle architecture and habituation to the eccentric pedaling task; Other: Pedaling at 15 rpm
- Eccentric pedalling group at 60 rpm (Experimental)
  Interventions: Other: Neuromuscular evaluation; Other: Assessment of aerobic capacity, muscle architecture and habituation to the eccentric pedaling task; Other: Pedaling at 60rpm
- Control (Active Comparator)
  Interventions: Other: Neuromuscular evaluation; Other: Assessment of aerobic capacity, muscle architecture and habituation to the eccentric pedaling task; Other: No pedaling, usual activity

INTERVENTIONS:
Other: Neuromuscular evaluation — Before and after training.
  Muscle function:
  * voluntary maximal isometric force of the knee extensors
  * evoked force in the knee extensors by double percutaneous electrical stimulation at 100 and 10 Hz
  * level of voluntary activation
  * voluntary maximum force in concentric and eccentric mode at an angular speed of 60°.s-1
  * squat jump and counter-movement jump
Other: Assessment of aerobic capacity, muscle architecture and habituation to the eccentric pedaling task — Before and after training.
  Cardiovascular-respiratory function:
  * Oxygen consumption during the incremental concentric pedaling test conducted to high effort perception.
  * heart rate during pedaling tasks
  Muscle architecture:
  - Pennation angle and thickness of vastus lateralis, rectus femoris, gastrocnemius medialis and lateralis muscles, before and after training.
  Familiarization with eccentric pedaling
Other: Pedaling at 15 rpm — 3 training sessions per week for 6 weeks
  Arms: Eccentric pedalling group at 15 rpm
Other: No pedaling, usual activity — Maintain usual physical activity and diet for a period of 6 weeks.
  Arms: Control
Other: Pedaling at 60rpm — 3 sessions per week of training for 6 weeks
  Arms: Eccentric pedalling group at 60 rpm

SUMMARY:
The recent appearance of ergocycles that can be used for eccentric pedaling (Cyclus type) has aroused a growing interest in the field of rehabilitation. The mechanical, metabolic, and cardiorespiratory characteristics of eccentric exercises make them an exercise of choice when the goal is to improve locomotor muscle function and exercise capacity. Despite its potential advantages, the optimal modalities of eccentric pedaling, in particular the choice of pedaling frequency, are still poorly understood, especially its effects on the neuromuscular system. Indeed, most training protocols impose a fixed pedaling power but with highly variable pedaling rates, ranging from 15 to 60 rpm (Besson et al., 2013; MacMillan et al., 2017). For a given pedaling power level (P), the choice of pedaling frequency (F) directly impacts the force torque (C) and thus the force applied to the pedals, since power is equal to the product of pedaling frequency and force torque (P = F.C). For frequencies varying from 15 to 60 rpm, the level of muscular tension during pedaling therefore varies from single to quadruple. These very large variations in force can influence the neuromuscular adaptations induced during a prolonged training period. For example, the use of low pedaling frequencies corresponding to high muscle tension could favor peripheral muscular adaptations (e.g. contractility) whereas higher pedaling frequencies could favor central (i.e. nervous) adaptations.

A better understanding of the neuromuscular adaptations induced by a period of eccentric pedaling at different cadences will allow for a more precise definition of training protocols for populations likely to undergo this type of training (e.g. elderly people, patients with heart failure).

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Subject capable of understanding simple commands and giving consent
* Subject (male or female) between 18 and 40 years of age.
* Subject able to do moderate physical activity

Exclusion Criteria:

* Person not affiliated to national health insurance.
* Physical disabilities affecting the lower limbs or the pelvis, and which may hinder or prevent the practice of exercise on an ergocycle, whether neurological (central or peripheral), arterial (in particular, arterial disease of the lower limbs with a systolic index < 0.6) or orthopedic (degenerative or inflammatory rheumatism).
* Person under legal protection (curatorship, guardianship)
* Person under court order (sauvegarde de justice)
* Pregnant, parturient or breastfeeding women
* Major unable to express consent
* Minor

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Maximum isometric force developed in the quadriceps | 6 weeks of training

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France